CLINICAL TRIAL: NCT03381339
Title: Powertoothbrushing for Treating Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Sunstar, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MarquetteU
Record Dates: First submitted 2017-12-18; First posted 2017-12-22 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Gingivitis
Keywords: power toothbrush, oscillating rotating
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: 3 month home use parallel-arm design to assess the efficacy of powered toothbrush use in the treatment of gingivitis in a moderate sized population, n=70.
Who Masked: Investigator
Masking Description: examiners will be unaware of which toothbrush has been assigned to each subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Powered toothbrush intervention (Experimental): Subjects will be provided an oscillating rotating powered toothbrush as the experimental intervention, and given written instructions on its proper use. Efficacy of overnight plaque reduction will be assessed at baseline and both gingivitis and plaque reduction will be assessed as change from baseline at 2, 4 and 12 weeks. Subjects will be given a standard fluoride toothpaste and asked to refrain from daily interproximal plaque control for the duration of the study.
  Interventions: Device: Oscillating rotating power toothbrush
- Manual toothbrush (No Intervention): Subjects will be provided a manual toothbrush as the control group and given written instructions on its proper use. Efficacy of overnight plaque reduction will be assessed at baseline and both gingivitis and plaque reduction will be assessed as change from baseline at 2, 4 and 12 weeks. Subjects will be given a standard fluoride toothpaste and asked to refrain from daily interproximal plaque control for the duration of the study.

INTERVENTIONS:
Device: Oscillating rotating power toothbrush — a battery powered oscillating rotating toothbrush will be used for twice daily regular home dental hygiene
  Other Names: powertoothbrush
  Arms: Powered toothbrush intervention

SUMMARY:
In this three-month interventional clinical trial for the treatment of gingivitis the investigators will assess the use of an oscillating-rotating powered toothbrush in comparison to the use of a manual toothbrush over 12-weeks in the absence of interproximal hygiene.

DETAILED DESCRIPTION:
In this single-masked, parallel-armed, interventional clinical trial for treatment of gingivitis the investigators will assess the use of an oscillating-rotating powered toothbrush in comparison to the use of a manual toothbrush over 12-weeks in the absence of interproximal hygiene. The primary outcome variable is the change from baseline in the Modified Gingival Index at 2, 4 and 12-weeks from Baseline. Secondary outcome variables include change from baseline in bleeding on probing as well as change from baseline in the Turesky Modification of the Quigley-Hein Plaque index measuring overnight plaque formation. There will also be an assessment of single use efficacy in reduction of overnight plaque levels at the baseline visit t

ELIGIBILITY:
Inclusion Criteria:

* A subject who meets all the following criteria will be eligible to enroll in this study.

  1. Age range 18 - 65 years
  2. Routine manual toothbrush user
  3. A Subject who agrees to use the assigned toothbrush as the only cleaning device for the study duration, refraining from daily interdental cleaning and/ or antiseptic mouthrinsing.
  4. Mild to moderate gingivitis as measured by A. Modified Gingival Index (MGI) average score of at least 1.2, and / or B. Bleeding on Probing (BOP) of at least 20% of all sites but not more than 50% of sites.
  5. Probing Pocket Depth (PPD) of 4 mm or lower
  6. At least 20 natural teeth - scoreable (crowns or bridgework are non-scoreable).

Exclusion Criteria:

* Any subject meeting one of the following criteria will not be included in the study.

  1. Daily user of interdental cleaning devices, such as floss, floss picks, toothpicks, interdental brush, water flossing device
  2. Regular user of antimicrobial mouthrinses within one week of entry into study
  3. Professional prophylaxis within one month of entry into the study
  4. Use of antibiotics within one month prior to the baseline exam
  5. Signs of moderate to severe periodontitis or caries, categorized as PPD of 5 mm of higher and attachment loss of 3 mm or higher
  6. Subjects with orthodontic bands and/or dental appliances.
  7. Participated in an oral care related study in the last 90 days prior to this study
  8. Pregnant or lactating women
  9. Patients with a history of significant cardiovascular disease, diabetes, cancer, AIDS, or other organ impairment that would preclude their participation in the study
  10. Acute/concurrent illness such as hepatitis, herpes simplex infections, influenza, etc.
  11. History of rheumatic fever, cardiovascular valvular disease, artificial joint replacement or kidney or liver disorders
  12. Chronic use of steroids; limited use of NSAID's (≤ 325 mg/day)
  13. Current Smoker (within the last 3 months)
  14. Other medical or dental conditions that would affect the study
  15. Inability to commit to all necessary study visits from baseline to 12 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Marquette University School of Dentistry, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medically healthy subjects between 18 and 65 years of age were recruited by posting flyers around the Milwaukee area.
Groups:
- Powered Toothbrush Intervention: Subjects will be provided an oscillating rotating powered toothbrush as the experimental intervention, and given written and professional oral instructions on its proper use at baseline 2 and 4 weeks. Efficacy of overnight plaque reduction will be assessed at baseline and both gingivitis and plaque reduction will be assessed as change from baseline at 2, 4 and 12 weeks. Subjects will be given a standard fluoride toothpaste and asked to refrain from daily interproximal plaque control for the duration of the study.
  Oscillating rotating power toothbrush: a battery powered oscillating rotating toothbrush will be used for twice daily regular home dental hygiene
- Manual Toothbrush: Subjects will be provided a manual toothbrush as the control group and given written and professional oral instructions on its proper use at baseline, 2 and 4 weeks. Efficacy of overnight plaque reduction will be assessed at baseline and both gingivitis and plaque reduction will be assessed as change from baseline at 2, 4 and 12 weeks. Subjects will be given a standard fluoride toothpaste and asked to refrain from daily interproximal plaque control for the duration of the study.
Period: Overall Study
Arm/Group | Powered Toothbrush Intervention | Manual Toothbrush
Started | 27 | 28
Completed (Subjects who completed all 12 weeks) | 23 | 24
Not Completed | 4 | 4
Not completed — Protocol Violation | 4 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Proportion of total number sites per patient. The score per gingival site is either 0 or 1 with 1 being bleeding after probing and 0 being no bleeding after probing. Since the unit of BOP measure is the patient and we made the measurement 4 times and each time we calculated full mouth score.
Units Other Than Participants: Bleeding Sites
Groups:
- Total: Total of all reporting groups
Arm/Group | Powered Toothbrush Intervention | Manual Toothbrush | Total
Number analyzed (Participants) | 23 | 24 | 47
Number analyzed (Bleeding Sites) | 3864 | 4032 | 7896
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.13 (8.42) | 25.75 (10.16) | 26.43 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 7 | 10 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 24 | 47
Bleeding on probing [Mean (Standard Deviation); unit: Average Bleeding Score] | 0.23 (0.08) | 0.27 (0.08) | 0.25 (0.09)

OUTCOME MEASURES:

1. Primary Outcome: Change in Gingivitis
Description: Baseline and 12 weeks post-baseline measures. Proportion of bleeding sites per patient was used as Full mouth BOP Score. The score for each site was either 1 for bleeding and 0 for no bleeding.
  Following is the full description of each outcome measure reported in the protocol.
  The Modified Gingival Index3 (MGI) will be measured on six sites - mesio-buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual - of all teeth using a 0-4 scale. Lower score no inflamation and higher severe inflammation.
  Dental plaque will be evaluated using the Lobene modification4 of the Turesky modification of the Quigley-Hein Plaque Index (PI)5. The score 0 to 5. Lower score means no plaque and higher score increasing plaque.Full-mouth Probing Pocket Depth (PPD) will be measured on the six locations of each tooth (mesial-buccal, buccal, distal-buccal, mesial-lingual, lingual, distal-lingual) using a periodontal probe.
Time Frame: 12 weeks post-baseline
Population: The analysis was on the number sites per patients. For BOP the score was for proportion of the bleeding sites. Similarly for MGI the score was full mouth average.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Powered Toothbrush Intervention | Manual Toothbrush
Number analyzed (Participants) | 23 | 24
score on a scale | 0.14 (0.07) | 0.19 (0.10)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Description: Pain
Groups:
- Powered Toothbrush Intervention: The patients were given power toothbrush with instructions to use
- Manual Toothbrush: The patients were given power manual toothbrush with instructions to use
Arm/Group | Powered Toothbrush Intervention | Manual Toothbrush
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03381339/Prot_SAP_ICF_000.pdf